CLINICAL TRIAL: NCT03879252
Title: Tolerance of Teeth Brushing During Prolonged Aplasia In Protected Unit
Brief Title: Tolerance of Teeth Brushing During Prolonged Aplasia
Acronym: UP-TIP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 49RC18_0147
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Aplasia
MeSH Terms: interventions — Mouthwashes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tooth brushing (Experimental)
  Interventions: Device: Toothbrush
- Mouthwash (Active Comparator)
  Interventions: Drug: Mouthwashes

INTERVENTIONS:
Device: Toothbrush — Brushing teeth three times a day (extra-soft toothbrush) with a 1.4% baking mouthwash solution.
  Arms: Tooth brushing
Drug: Mouthwashes — Mouthwashes three times a day with a 1.4% baking mouthwash solution.
  Arms: Mouthwash

SUMMARY:
It is currently not allowed for patients with prolonged aplasia, following intensive chemotherapy, to brush teeth due to the risk of damaging the oral mucosa with risk of haemorrhage and infectious entrance door. Mouthwash is currently prescribed to prevent these complications. Many patients, however, ask to brush their teeth for greater comfort and a feeling of well-being.

Some haematology services allow tooth brushing while others prohibit tooth brushing without study.

Investigators wanted to conduct a study to assess the feasibility, the safety of tooth brushing for aplastic patient comfort, hemopathy and/or chemotherapies causing mucous membrane alteration that increases infectious risk and the risk of gingivorragia.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized Patients in protected area of the Blood Disease Service with predictable prolonged aplasia and risk of mucite
* Acute myeloblastic leukemia undergoing induction or consolidation treatment
* Acute lymphoblastic leukemia under induction treatment
* Patients affiliated or beneficiaries of a social security
* Written inform consent

Exclusion Criteria:

* Patients with removable complete dentures
* Constitutional disorder of coagulation
* Hematopoietic stem cell allogreffe
* Therapeutic intensification with autograft of haematopoietic stem cells
* Patient unable to provide oral care alone (brushing teeth or mouthwash)
* Already included in the study
* Pregnant women, lactating mothers
* Persons deprived of liberty by an administrative or judicial decision
* Persons undergoing psychiatric care under duress
* Adults who are subject to a legal or non-state protection measure to express their consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Highest score obtained at the OAG (Oral Assessment Guide) scale during the observation period | 1 month
  Assess the effect of the "teeth brushing" versus "mouth bath" strategy on the oral condition of patients hospitalized in the protected area of the Blood Disease Service with predictable prolonged aplasia and risk of mucite

SECONDARY OUTCOMES:
Number of septicemia | 1 month
  Estimate the effect of the strategy in terms of Infectious risks
Incidence of intra-oral hemorrhage | 1 month
  Estimate the effect of the strategy in terms of Hemorrhagic risk
Number of days with intra-oral hemorrhage | 1 month
  Estimate the effect of the strategy in terms of Hemorrhagic risk
Number of days with fever | 1 month
  Estimate the effect of the strategy in terms of Infectious risks
Incidence of bacterial infections during hospitalization | 1 month
  Estimate the effect of the strategy in terms of Infectious risks
Incidence of fungal infections during hospitalization | 1 month
  Estimate the effect of the strategy in terms of appearance of mucite
Percentage of patients receiving morphinics during hospitalization | 1 month
  Estimate the effect of the strategy in terms of pain
Number of days with morphinic treatment | 1 month
  Estimate the effect of the strategy in terms of pain
Percentage of patients receiving parenteral nutrition during hospitalization | 1 month
  Estimate the effect of the strategy in terms of patient's tolerance to oral care
Number of days with parenteral nutrition | 1 month
  Estimate the effect of the strategy in terms of patient's tolerance to oral care
Percentage of patients who had to discontinue treatment on medical advice | 1 month
  Estimate the effect of the strategy in terms of patient's tolerance to oral care

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Angers, Angers, France

IPD SHARING:
Plan to Share IPD: No